CLINICAL TRIAL: NCT01297465
Title: A Phase IIIB, Multicentre, Multinational, Randomized, Open-label Trial to Compare the Efficacy and Safety of Ovarian Stimulation With GONAL-f® Day 1 to Day 5 Followed by Pergoveris® Starting Day 6 to Pergoveris® Starting Day 1 in Women Between 36 and 40 Years of Age Undergoing Assisted Reproductive Technique (ART)
Brief Title: PERgoveriS In Stratified Treatment for Assisted Reproductive Technique
Acronym: PERSIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A., Geneva (Industry); Merck A/S, Denmark (Industry); Merck OY, Finland (Industry); Merck Serono S.A.S, France (Industry); Merck Serono GmbH, Germany (Industry); Merck A.E., Greece (Industry); Merck B.V., Netherlands (Industry); Merck SP. Z.O.O., Poland (Industry); Merck Serono S.P.A., Italy (Industry); Merck Services U.K. Ltd, UK (Industry); LLC Merck, Russia (Industry); Merck spol. s r.o., Slovakia (Industry); Merck Pharma, K.S., Slovakia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200061-504; 2010-023534-23 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Assisted Reproductive Techniques; Reproductive Technology, Assisted
Keywords: Ovulation Induction; Ovarian Stimulation; Reproductive Technique, Assisted; Assisted Reproductive Technics; Assisted Reproductive Technique; Reproductive Technology, Assisted
MeSH Terms: conditions — Helping Behavior | interventions — follitropin alfa; pergoveris; Chorionic Gonadotropin; Ovidrel

ARMS (2):
- Gonal-f® Plus Pergoveris® (Active Comparator)
  Interventions: Drug: Gonal-f®; Drug: Pergoveris®; Drug: Recombinant human chorionic gonadotropin (r-hCG)
- Pergoveris® (Experimental)
  Interventions: Drug: Pergoveris®; Drug: Recombinant human chorionic gonadotropin (r-hCG)

INTERVENTIONS:
Drug: Gonal-f® — Gonal-f® (follitropin alfa) 300 International Unit (IU) will be administered subcutaneously once daily from stimulation day 1 (S1) to stimulation day 5 (S5).
  Other Names: Follitropin alfa
  Arms: Gonal-f® Plus Pergoveris®
Drug: Pergoveris® — Pergoveris® (follitropin alfa and lutropin alfa) 300 IU will be administered subcutaneously starting from S6 until recombinant human chorionic gonadotropin (r-hCG) administration day (at least 1 follicles >= 18 mm). The dose of Pergoveris® was adjusted based upon the participant's ovarian response and according to the site's standard practice.
  Arms: Gonal-f® Plus Pergoveris®
Drug: Pergoveris® — Pergoveris® (follitropin alfa and lutropin alfa) 300 IU will be administered subcutaneously once daily from S1 until r-hCG administration day (at least 1 follicles >= 18 mm). The dose of Pergoveris® was adjusted starting from S6 based upon the participant's ovarian response and according to the site's standard practice.
  Arms: Pergoveris®
Drug: Recombinant human chorionic gonadotropin (r-hCG) — 250 microgram of r-hCG will be administered once subcutaneously on r-hCG day (at least 1 follicles >= 18 mm).
  Other Names: Ovidrel®; Ovitrelle®

SUMMARY:
This is a multicenter, multi-national, randomized, open-label comparative trial. After screening, the subjects will start down-regulation treatment on Day 21-22 of the cycle. Down-regulation treatment will start within 2 months following the screening visit. The routine long luteal phase protocol for gonadotropin-releasing hormone (GnRH) agonist treatment will be followed. Once down-regulation has been confirmed, a pregnancy test will be performed just before randomization and start of recombinant human follicle-stimulating hormone (r-hFSH) treatment to rule out any pre-existing pregnancy. If the result is negative, the subject will be randomly assigned to one of the two treatment arms of the trial:

* GONAL-f®: (Liquid Pen; 300 international unit [IU] of per day) stimulation Day 1-5 followed by Pergoveris® (vial/powder, 300 IU per day) from stimulation Day 6 and until required recombinant human chorionic hormone (r-hCG) criterion is met. The dose can be adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.
* Pergoveris®: (vial/powder, 300 IU per day) from stimulation Day 1 and until required r-hCG criterion is met. The dose can be adjusted from stimulation Day 6 (increased or decreased) based upon the subject's ovarian response and according to the center's standard practice.

Randomization across the two treatment arms will be kept balanced in a 1:1 ratio. Follicular development will be monitored according to the center's standard practice by ultrasound (US) and/or estradiol (E2) levels, until the protocol r-hCG requirement is met (i.e., at least one follicle greater than or equal to [>=] 18 millimeter [mm] and two follicles >=16 mm). After this, a single injection of r-hCG will be administered in order to induce final oocyte maturation.

At a time of 34-38 hours after r-hCG administration, oocytes will be recovered vaginally under US monitoring. Oocytes will then be fertilized in vitro and embryos replaced 2-5 days after oocyte recovery. Ovum pick up (OPU), in vitro fertilization (IVF), embryo transfer (ET) and luteal support will be performed as per center's standard practice.

A post-treatment safety visit will be performed for all subjects who received r-hCG (pregnant and non- pregnant) on Day 15-20 post-hCG. For subjects who have withdrawn from treatment (i.e. after starting Pergoveris® or Gonal-f® but before hCG is given) this visit will take place 20-30 days after their first Pergoveris® or Gonal-f® treatment injection (excluding pregnancy testing).

ELIGIBILITY:
Inclusion Criteria:

* Be a female subject justifying an in vitro fertilization and embryo transfer (IVF/ET) treatment
* Be between her 36th and 40th birthday (both included) at the time of the randomization visit
* Have early follicular phase (Day 2-4) serum level of basal follicle stimulating hormone (FSH less than or equal to (=<)12 IU/L) measured in the center's local laboratory during the screening period (that is within 2 months prior to down-regulation start)
* A body mass index (BMI) less than (<) 30 kilogram per square meter (kg/m^2)
* Have a regular spontaneous ovulatory menstrual cycle between 21 and 35 days in length
* Be willing and able to comply with the protocol for the duration of the trial
* Have given written informed consent, prior to any trial-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to her future medical care
* Have a male partner with semen analysis within the past 6 months prior to randomization considered adequate to proceed with regular insemination or intracytoplasmic sperm injection (ICSI) according to the center's standard practice. If these criteria are not met, the subject can only be entered if donor sperm will be used
* Other protocol specified inclusion criteria could also apply.

Exclusion Criteria:

* Had >= 2 previous ART cycles with a poor response to gonadotrophin stimulation defined as =< 6 mature follicles and/or =<4 oocytes collected in any previous IVF cycle or previous cycles with a hyper response defined as >= 25 oocytes retrieved
* Any medical condition, which in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug. In case of doubt, the subject in question should be discussed with Merck Serono's medical responsible
* Had previous severe ovarian Hyperstimulation Syndrome (OHSS)
* Polycystic ovary syndrome (PCOS; Rotterdam criteria) to reduce the risk of the occurrence of OHSS
* Any contraindication to being pregnant and/or carrying a pregnancy to term
* History of 3 or more miscarriages (early or late miscarriages) due to any cause
* A clinically significant systemic disease
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus in the trial subject or her male partner
* Known allergy or hypersensitivity to human gonadotrophin preparations
* Entered previously into this trial or simultaneous participation in another clinical trial.
* Pregnancy and lactation period
* Participation in another clinical trial within the past 30 days
* Other protocol specified inclusion criteria could also apply.

Ages: 36 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Longobardi, MD, Study Director — Merck Serono S.P.A., Italy
Locations (23):
- Denmark (2):
  - Research Site, Dronninglund
  - Research Site, Fredericia
- Research Site, Helsinki, Finland
- France (5):
  - Research Site, Bondy
  - Research Site, Bruges
  - Research Site, Clamart
  - Research Site, Thenon
  - Research Site, Villeurbanne
- Germany (2):
  - Research Site, Berlin
  - Research Site, Halle
- Greece (3):
  - Research Site, Heraklion, Crete
  - Research Site, Pylaia, Thessaloniki
  - Research Site, Athens
- Italy (3):
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Torino
- Research Site, Zwolle, Netherlands
- Research Site, Warsaw, Poland
- Russia (2):
  - Research Site, Moscow
  - Research Site, Samara
- Research Site, Bratislava, Slovakia
- United Kingdom (2):
  - Research Site, London
  - Research Site, Swansea

REFERENCES:
- [Result] H Behre, C Howles, S Longobardi. Luteinizing hormone supplementation from Day 1 versus 6 of ovarian stimulation in women aged 36-40 years: results from an open-label, randomized, multicentre, multinational trial. Human Reproduction. 2013;28(suppl 1)
- [Result] Behre HM, Howles CM, Longobardi S; PERSIST Study Investigators. Randomized trial comparing luteinizing hormone supplementation timing strategies in older women undergoing ovarian stimulation. Reprod Biomed Online. 2015 Sep;31(3):339-46. doi: 10.1016/j.rbmo.2015.06.002. Epub 2015 Jun 15. PMID 26194884

RESULTS

PARTICIPANT FLOW:
Groups:
- Gonal-f® Plus Pergoveris®: Gonal-f® (follitropin alfa) 300 International Unit (IU) was administered subcutaneously once daily from stimulation day 1 (S1) to stimulation day 5 (S5) followed by subsequent daily administration of Pergoveris® (follitropin alfa and lutropin alfa) 300 IU subcutaneously starting from S6 until recombinant human chorionic gonadotropin (r-hCG) (Ovidrel®/Ovitrelle®) administration day (at least 1 follicles greater than or equal to (>=) 18 millimeter [mm]). On r-hCG day, 250 microgram of r-hCG was administered once subcutaneously. The dose of Pergoveris® was adjusted based upon the participant's ovarian response and according to the site's standard practice.
- Pergoveris®: Pergoveris® (follitropin alfa and lutropin alfa) 300 IU was administered subcutaneously once daily from S1 until r-hCG administration day (at least 1 follicles >= 18 mm). On r-hCG (Ovidrel®/Ovitrelle®) day, 250 microgram of r-hCG was administered once subcutaneously. The dose of Pergoveris® was adjusted starting from S6 based upon the participant's ovarian response and according to the site's standard practice.
Period: Overall Study
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Started | 99 | 103
Completed | 91 | 93
Not Completed | 8 | 10
Not completed — Lack of Ovarian Response | 1 | 1
Not completed — Ovarian hyperstimulation syndrome risk | 0 | 1
Not completed — No Oocytes Retrieved | 1 | 1
Not completed — Poor oocyte quality | 0 | 1
Not completed — No Fertilization | 6 | 4
Not completed — All Embryos Discarded | 0 | 1
Not completed — Intention to Freeze all Embryos | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all the randomized participants who had received at least 1 dose of Pergoveris® or Gonal-f®.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris® | Total
Number analyzed (Participants) | 99 | 103 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (1.16) | 37.4 (1.14) | 37.5 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 103 | 202
  Male | 0 | 0 | 0
Race [Number; unit: participants]
  Black | 4 | 3 | 7
  Asian | 4 | 6 | 10
  Other | 2 | 2 | 4
  White | 89 | 92 | 181
Height [Mean (Standard Deviation); unit: centimeter] | 166.1 (6.49) | 166.3 (6.47) | 166.2 (6.46)
Weight [Mean (Standard Deviation); unit: kilogram] | 64.81 (10.364) | 65.82 (8.923) | 65.33 (9.645)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Oocytes Retrieved
Description: The total number of oocytes retrieved per reporting group on the day of ovum pick-up (OPU) (34-38 hours post r-hCG day) was calculated. Oocyte retrieval is a technique used in in-vitro fertilization (IVF) in order to remove oocytes from the ovary of the female participant, enabling fertilization outside the body.
Time Frame: OPU day (34-38 hours post r-hCG day [end of stimulation cycle {approximately 11 days}])
Population: Modified intention-to-treat (Mod-ITT) population included all the randomized participants who had received at least one dose of GONAL-f® or Pergoveris®, and completed the primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 98 | 101
oocytes | 10.9 (6.5) | 9.7 (6.9)
Statistical Analysis 1: Comparison: Gonal-f® Plus Pergoveris® vs Pergoveris®; The null hypothesis was that the difference between the mean number of oocytes is less than (-3) or greater than (+3) between the two treatment arm. The alternate hypothesis was that the difference is between (-3) and (+3). The study had 80% power to show that the group randomized to Pergoveris® has an absolute difference of no more than 3 oocytes retrieved in comparison to the group randomized to GONAL-f®/Pergoveris®; Test type: Superiority or Other; ANOVA; ANOVA model adjusted for treatment and country; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-3.15 to 0.59], Standard Error of Mean 0.947 — The primary efficacy variable was to be analyzed using an analysis of variance (ANOVA) model, adjusted for treatment and country

2. Secondary Outcome: Total Dose and Mean Daily Dose of Follicle Stimulating Hormone (FSH)
Time Frame: Day 1 up to r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Safety Population included all the randomized participants who had received at least 1 dose of Pergoveris® or Gonal-f®.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 99 | 103
IU
  Total Dose | 3292 (851) | 3321 (850)
  Mean Daily Dose | 307 (43) | 311 (41)

3. Secondary Outcome: Total Number of Stimulation Treatment Days
Time Frame: Day 1 up to r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Safety Population included all the randomized participants who had received at least 1 dose of Pergoveris® or Gonal-f®.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 99 | 103
days | 10.6 (1.6) | 10.6 (1.7)

4. Secondary Outcome: Implantation Rate
Description: Implantation rate per reporting group was measured as the number of fetal sacs observed, divided by the number of embryos transferred multiplied by 100.
Time Frame: Days 35-42 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Mod-ITT population included all the randomized participants who had received at least one dose of GONAL-f® or Pergoveris®, and completed the primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: percent sacs per embryo
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 90 | 93
percent sacs per embryo | 13.3 (29.1) | 24.7 (36.1)

5. Secondary Outcome: Number of Fetal Sacs With Activity
Description: Number of fetal sacs with activity was evaluated by ultrasound scan
Time Frame: Days 35-42 post r-hCG day [end of stimulation cycle {approximately 11 days}])
Population: Mod-ITT population included all the randomized participants who had received at least one dose of GONAL-f® or Pergoveris®, and completed the primary efficacy assessment."N" (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: fetal sacs
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 18 | 35
fetal sacs | 1.4 (0.5) | 1.2 (0.4)

6. Secondary Outcome: Number of Fetal Hearts With Activity
Description: Number of fetal hearts with activity was evaluated by ultrasound scan
Time Frame: Days 35-42 post r-hCG day [end of stimulation cycle {approximately 11 days}])
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: fetal hearts
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 17 | 32
fetal hearts | 1.4 (0.5) | 1.3 (0.5)

7. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy was defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy. Clinical pregnancy rate was reported as total clinical pregnancy rate, clinical pregnancy rate per cycle started and per embryo transfer [ET]).
Time Frame: Days 35-42 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Mod-ITT population included all the randomized participants who had received at least one dose of GONAL-f® or Pergoveris®, and had completed the primary efficacy assessment. "N" signifies those participants who had their ET in study treatment cycle. "n" signifies those participants who were evaluated for this measure in specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 97 | 101
percentage of participants
  Total clinical pregnancy rate (n=97, 101) | 17.5 | 31.7
  Clinical pregnancy rate per cycle (n=97, 101) | 17.5 | 31.7
  Clinical pregnancy rate per ET (n=90, 93) | 18.9 | 34.4

8. Secondary Outcome: Number of Participants With Cancelled Cycles Due to Excessive or Insufficient Ovarian Response to Treatment
Description: An excessive ovarian response: greater than or equal to 25 oocytes which could put the participant at risk of OHSS; An insufficient ovarian response: defined as 3 or less follicles of greater than or equal to 12 millimeter developing following at least 7 days of treatment.
Time Frame: S1 until Day 15-20 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Safety Population included all the randomized participants who had received at least 1 dose of Pergoveris® or Gonal-f®.
Measure: Number; unit: participants
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 99 | 103
participants
  Insufficient ovarian response | 1 | 1
  Excessive ovarian response | 0 | 1

9. Secondary Outcome: Biochemical Pregnancies Rate
Description: Biochemical pregnancy was defined as the pregnancy diagnosed only by the detection of human chorionic gonadotropin (hCG) in serum or urine and that does not develop into a clinical pregnancy. Participants with beta- hCG concentration greater than 10 international units per liter (IU/L) were considered as biochemical pregnant.
Time Frame: Days 15-20 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Mod-ITT population included all the randomized participants who had received at least one dose of GONAL-f® or Pergoveris®, and completed the primary efficacy assessment. . "N" (number of participants analyzed) signifies those participants who had their embryo transfer in study treatment cycle.
Measure: Number; unit: participants
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 97 | 101
participants | 23 | 41

10. Secondary Outcome: Number of Participants With Multiple Pregnancies
Description: Multiple pregnancy was defined as the existence of more than one fetal sac with fetal heart activity.
Time Frame: Days 35-42 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Mod-ITT population included all the randomized participants who had received at least one dose of GONAL-f® or Pergoveris®, and completed the primary efficacy assessment. "N" (number of participants analyzed) signifies those participants who had their embryo transfer in study treatment cycle.
Measure: Number; unit: participants
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 97 | 101
participants | 6 | 8

11. Secondary Outcome: Number of Participants With Early and Late Ovarian Hyper Stimulation Syndrome (OHSS)
Description: Ovarian Hyper Stimulation Syndrome (OHSS) is a syndrome which can manifest with enlarged ovaries, advanced ascites with increased vascular permeability, pleural fluid accumulation, hemoconcentration, and increased blood clotting. Early OHSS was defined as the onset of OHSS occurring within 9 days after oocyte retrieval and late OHSS was defined as the onset of OHSS occurring on or after day 10 from oocyte retrieval.
Time Frame: Days 15-20 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Safety Population included all the randomized participants who had received at least 1 dose of Pergoveris® or Gonal-f®.
Measure: Number; unit: participants
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 99 | 103
participants
  Early Ovarian hyperstimulation syndrome | 4 | 1
  Late Ovarian hyperstimulation syndrome | 0 | 1

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Day 1 up to days 15-20 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Safety Population included all the randomized participants who had received at least 1 dose of Pergoveris® or Gonal-f®.
Measure: Number; unit: participants
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 99 | 103
participants | 26 | 23

13. Secondary Outcome: Systolic and Diastolic Arterial Blood Pressure Assessments
Time Frame: Days 15-20 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: Safety Population included all the randomized participants who had received at least 1 dose of Pergoveris® or Gonal-f®. ."N" (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter of mercury ( mm Hg)
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 93 | 99
millimeter of mercury ( mm Hg)
  Systolic Blood Pressure | 118.9 (12.8) | 121.2 (14.8)
  Diastolic Blood Pressure | 74.8 (9.8) | 76.8 (9.5)

14. Secondary Outcome: Heart Rate Assessments
Time Frame: Days 15-20 post r-hCG day (end of stimulation cycle [approximately 11 days])
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Number analyzed (Participants) | 93 | 99
beats per minute (bpm) | 75.7 (10.5) | 76.5 (10)

ADVERSE EVENTS:
Time Frame: Days 15-20 post r-hCG day (end of stimulation cycle [approximately 11 days])
Arm/Group | Gonal-f® Plus Pergoveris® | Pergoveris®
Serious Adverse Events (participants affected / at risk) | 2/99 | 0/103
Other Adverse Events (participants affected / at risk) | 31/99 | 32/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gonal-f® Plus Pergoveris® (N=99) | Pergoveris® (N=103)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gonal-f® Plus Pergoveris® (N=99) | Pergoveris® (N=103)
Headache (Nervous system disorders) | 14 | 13
Somnolence (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Lip pruritus (Gastrointestinal disorders) | 1 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 3 | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 2
Adnexa uteri pain (Reproductive system and breast disorders) | 2 | 2
Breast pain (Reproductive system and breast disorders) | 1 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 6
Oral herpes (Infections and infestations) | 1 | 1
Escherichia vaginitis (Infections and infestations) | 1 | 0
Eye infection viral (Infections and infestations) | 0 | 1
Vaginitis bacterial (Infections and infestations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Injection site induration (General disorders) | 0 | 1
Waist circumference increased (Investigations) | 2 | 0
Oestradiol increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Hot flush (Vascular disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Myopia (Eye disorders) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less